CLINICAL TRIAL: NCT00180440
Title: INcidence Free SUrvival Before and After ICD Replacement
Brief Title: INSURE: INcidence Free SUrvival Before and After Implantable Cardioverter Defibrillator (ICD) Replacement
Status: Completed | Type: Observational
Sponsor: Guidant Corporation (Industry)
Responsible Party: Andrea Ungefehr, Guidant Germany a Boston Scientific company
Other Study IDs: INSURE 1.3
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2009-03-26 (Estimated); Status verified 2009-03

CONDITIONS: Ventricular Fibrillation
MeSH Terms: conditions — Ventricular Fibrillation | interventions — Defibrillators, Implantable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Device: ICD — all models of Guidant/Bsc ICD's
  Other Names: implantable defibrillator

SUMMARY:
The INSURE trial is a multi-center, prospective trial to collect information about adequate ICD therapies in ICD patients before and after their first elective ICD replacement.

DETAILED DESCRIPTION:
The INSURE trial is a multi-center, prospective trial to collect information about adequate ICD therapies in ICD patients before & after their first elective ICD replacement. For this purpose all consecutive ICD patients will be included in the study, whose first implanted device is replaced due to ICD battery depletion (i.e. arrival at battery indicator ERI). ICD replacements due to other reasons can be included if duration of first ICD implantation was > 3 years. All patients included in the trial are regularly followed up until delivery of their first adequate ICD therapy. The collected data shall provide statistically valid information about the risk to patients who never have experienced adequate ICD therapy before the ICD replacement investigated in this study. In the future, these statistical risk data can give additional information to implanting physicians, such as whether an ICD replacement can eventually be omitted in those patients who are at very low risk for the occurrence of ICD therapies. All actually available GUIDANT ICDs with CE certificate can be implanted in this trial.

ELIGIBILITY:
Inclusion Criteria:

* All elective ICD replacements due to battery depletion of the first ICD being implanted in the patient

Exclusion Criteria:

* Non-availability to regular follow-up
* Age < 18 years
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all patients who are considered for ICD replacement due to normal battery depletion
Sampling Method: Non-Probability Sample
Enrollment: 528 (Estimated)
Dates: Start 2002-07; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johannes Sperzel, MD, Principal Investigator — Kerckhoff Klinik
Locations (1):
- IKKF, Insitut für Klinisch-kardiovaskuläre Forschung, München, Germany